CLINICAL TRIAL: NCT04360980
Title: Effects of Standard Protocol Therapy With or Without Colchicine in Covid-19 Infection: A Randomized Double Blind Clinical Trial
Brief Title: The Effects of Standard Protocol With or Without Colchicine in Covid-19 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nooshin dalili, Principal Investigator, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBMU.IR.REC.165423
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): 40 RT-PCR positive COVID-19 patients without hypoxemia administered Colchicine plus standard treatment
  Interventions: Drug: Colchicine Tablets
- Standard treatment (No Intervention): 40 RT-PCR positive COVID-19 patients without hypoxemia receiving vitamin C 3grams daily , 400 mg Tiamine, Selenium , Omega-3 500 mg daily, Vit A , Vit D, Azithromycine, Ceftriaxone, Kaletra 400 BID 10 days

INTERVENTIONS:
Drug: Colchicine Tablets — 1.5 mg loading then 0.5 mg BID P.O
  Other Names: Colchicine
  Arms: Intervention

SUMMARY:
Based on data regarding the effect of colchicine on the modulation of immune system and decreasing cytokine release and inflammation the question arises whether colchicine, administered in a relatively low dose, could potentially have an effect on COVID-19 Polymerase chain reaction(PCR) positive patients .

DETAILED DESCRIPTION:
80 Patients with positive nasopharyngeal swab PCR for COVID-19 which were not hypoxic but showed computed tomography involvement compatible with COVID-19 admitted in ward (not in Intensive care unit) included and randomized in to two groups. All patients received standard treatment protocol including essential minerals, vitamins as antioxidants, antibiotics and Kaletra while in one randomly assigned group colchicine would be added.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old with nasopharyngeal swab confirmed COVID-19 PCR, CT involvement compatible with COVID, Fever and Dyspnea without hypoxemia.

Exclusion Criteria:

* Patient who is not willing to enter in study
* Known hypersensitivity to colchicine
* Hepatic failure
* Renal failure with eGFR<20 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
CRPxN/R ratio change | 2 weeks
  increasing inflammatory status
Clinical deterioration by the WHO definition | 2 weeks
  including change in fever or O2 Saturation
PCR Viral Load | 2 weeks
  change in RT-PCR
CT severity involvement index | 2weeks
  change in CT involvement

SECONDARY OUTCOMES:
LDH change | 2 weeks
  change in LDH

CONTACTS AND LOCATIONS:
Overall Officials: SBMU, Principal Investigator — CKDRC,SBMU
Locations (2):
- Iran (2):
  - SBMU, Tehran
  - Nooshin Dalili, Tehran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dalili N, Kashefizadeh A, Nafar M, Poorrezagholi F, Firouzan A, Samadian F, Samavat S, Ziaie S, Fatemizadeh S. Adding Colchicine to the Antiretroviral Medication - Lopinavir/Ritonavir (Kaletra) in Hospitalized Patients with Non-Severe Covid-19 Pneumonia: A Structured Summary of a Study Protocol for a Randomized Controlled Trial. Trials. 2020 Jun 5;21(1):489. doi: 10.1186/s13063-020-04455-3. PMID 32503620